CLINICAL TRIAL: NCT03779113
Title: A Phase I, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HMPL-523 in Patients With Relapsed or Refractory Lymphoma
Brief Title: An Open-label, Dose Escalation Trial to Evaluate the Safety and Pharmacokinetics of HMPL-523 in Patients With Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-523-00US1
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Non Hodgkin Lymphoma
Keywords: lymphoma; chronic lymphocytic leukemia; Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients to received study drug (HMPL-523)
  Interventions: Drug: HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — Oral HMPL-523

SUMMARY:
This is a Phase I, open-label, multicenter study of HMPL-523 administered orally to patients with relapsed or refractory lymphoma who have exhausted approved therapy options. This study consists of a dose escalation stage (Stage1) and a dose expansion stage (Stage 2).

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicenter study of HMPL-523 administered orally to patients with relapsed or refractory lymphoma who have exhausted approved therapy options. This study consists of a dose escalation stage (Stage1) and a dose expansion stage (Stage 2).

Dose Escalation Stage (Stage 1)

Dosing will begin at 100 mg once daily (QD). A cycle of study treatment will be defined as 28 days of continuous dosing. The modified 3+3 design will be applied for dose escalation and MTD determination to limit the number of patients exposed to potentially ineffective or unsafe doses. The study will enroll 1 patient and the patient will be treated for a 28-day cycle in the initial dose cohort. If there is no Dose Limiting Toxicity (DLT) and no more than 2 treatment-emergent adverse events (TEAEs) of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 in the first treatment cycle, the study will be escalated to the next dose cohort and continue with the standard 3+3 design. Otherwise, the trial will revert to a standard 3+3 design from the initial dose cohort. A minimum of 3 patients will be enrolled and observed for toxicity in each successive dose cohort after the initial dose cohort. If the 3 patients initially enrolled in a given dose cohort complete the DLT assessment window (Cycle 1, Days 1-28) without experiencing a DLT, 3 patients will be enrolled at the next higher dose level. If 2 or more of the initial 3 patients enrolled at any dose level experience a DLT during the DLT assessment window, the dose escalation will be halted. If 1 of the initial 3 patients enrolled at any dose level experiences a DLT during the DLT assessment window, additional patients will be enrolled at that dose level for a minimum of 6 evaluable patients for DLT. If a DLT is observed in 1 of the 6 valuable patients at this dose level, dose escalation will proceed to the next pre- defined dose level. If DLTs are observed in 2 or more of the 6 evaluable patients at a given dose level, the dose escalation will be halted. If the dose escalation is completed due to 2 or more DLTs at a dose level and that dose level is ≥50% higher than the previous dose level, then an intermediate dose level may be evaluated for toxicity in the same manner as described above. If the dose level is <50% higher than the previous dose level, in which only 3 DLT evaluable patients were enrolled, 3 additional patients will be enrolled at that dose level to comprise 6 DLT evaluable patients.

The proposed dose escalation scheme comprises Cohorts 1 to 5 with dosing levels of 100 mg QD, 200 mg QD, 400 mg QD, 600 mg QD and 800 mg QD, respectively. The need for dose escalation beyond 800 mg QD, the specific dose to be tested and the potential for twice-daily (BID) dosing will be evaluated jointly by investigators and the sponsor based on the cumulative clinical safety, pharmacokinetic, and preliminary efficacy data. Safety monitoring and evaluation of dose escalation will be carried out by the Safety Review Committee, which will be comprised of the sponsor's study team members (including medical monitor, safety monitor and and Pharmacokinetic scientist) and the site principal investigators. The adverse event profile and serum concentration of HMPL-523 data will be evaluated to determine whether it is safe to continue the assigned HMPL-523 dose for dose escalation or whether the dose should be de-escalated to the lower dose level.

Dose Expansion Stage (Stage 2)

The adverse event profile, serum concentration, and preliminary anti-tumor activity of HMPL-523 at the maximum tolerated dose(MTD)/recommended phase 2 dose(RP2D) will be further evaluated in approximately 50 patients with relapsed or refractory indolent B-cell non-Hodgkin's lymphomas. The tumor types of the dose expansion stage are restricted to:

* 10 patients with chronic lymphocytic leukemia/small lymphocytic lymphoma
* 20 patients with chronic lymphocytic leukemia/small lymphocytic lymphoma post-BTK exposure
* 10 patients with mantle cell lymphoma
* 20 patients with follicular lymphoma (Grade 1-3a)
* 10 patients with marginal zone lymphoma
* 10 patients with waldenström's macroglobulinemia/lymphoplasmacytic lymphoma
* 10 patients with peripheral T- cell lymphoma
* 10 patients with cutaneous B-cell lymphoma
* 10 patients with hodgkin lymphoma

Patients will receive HMPL-523 at the MTD/RP2D for continuous 28-day treatment cycles until disease progression, death, intolerable toxicity, at investigator's discretion that the patient can no longer benefit from the study treatment, patient withdrawal from the study, or the end of study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to be eligible for study entry:

1. Signed informed consent form (ICF).
2. Age ≥18 years.
3. ECOG performance status of 0 or 1.
4. Histologically confirmed lymphoma, including Hodgkin's lymphoma and non-Hodgkin's lymphoma. In the dose expansion stage, the tumor types may be restricted to any or all of the following tumor types. There may be approximately 10 patients in each cohort depending on response signals suggesting efficacy, except for 2 identified cohorts with approximately 20 patients per cohort: relapsed or refractory CLL/SLL, CLL/SLL post-BTK exposure (n=20), MCL, FL (Grade 1-3a) (n=20), MZL, WM/LPL, PTCL,CBCL, and/or HL
5. Patients with relapsed or refractory lymphoma who have exhausted all approved therapy options.
6. In the dose expansion stage, patients must have measurable disease for an objective response assessment, except for patients with CLL and WM/LPL
7. Availability of tumor sample for patients in dose expansion cohorts: This may be an archival tissue sample obtained after most recent therapy or a fresh biopsy; if tumor sample is not available, the Sponsor may waive the requirement after discussion
8. Expected survival of more than 24 weeks as determined by the investigator.
9. Male patients must agree to use a condom and female patients of childbearing potential must agree to use highly effective contraceptive measures for 30 days after the last dose of study drug. These include as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, and transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, and implantable), intrauterine contraceptive device, intrauterine hormone release system, bilateral tubal occlusion, or a vasectomized partner, provided that male partner is the sole sexual partner of the female patient. Postmenopausal females (women who have not had menses for at least 1 year without an alternative medical cause) are exempt from this criterion.

Exclusion Criteria

1. Patients with primary central nervous system (CNS) lymphoma.
2. Any of the following laboratory abnormalities: Absolute neutrophil count<1.0×10^9/L, Hemoglobin <80 g/L, Platelets <50×10^9/L
3. Inadequate organ function, defined by the following: Total bilirubin >1.5 times the upper limit of normal (× ULN), aspartate aminotransferase and/or alanine aminotransferase >2.5 × ULN, Estimated Creatinine Clearance (CrCl) per Cockcroft-Gault [Dose Escalation portion of trial (Stage 1) CrCl < 40 mL/min, Dose Expansion portion of trial (Stage 2) CrCl < 30 mL/min], Serum amylase or lipase >ULN, International normalized ratio >1.5 × ULN, or activated partial thromboplastin time >1.5 × ULN
4. Patients with clinically detectable second primary malignant tumors at enrollment or other malignant tumors within the last 2 years (with the exception of radically treated basal cell or squamous cell carcinoma of the skin, in situ cervix, or in situ breast cancer).
5. Any anticancer therapy, including chemotherapy, hormonal therapy, biologic therapy, vaccine, or radiotherapy within 3 weeks prior to the initiation of study treatment.
6. Herbal therapy within 1 week prior to the initiation of study treatment.
7. Prior use of any anti-cancer vaccine
8. Prior treatment with any spleen tyrosine kinase (SYK) inhibitors (eg, fostamatinib)
9. Prior administration of radioimmunotherapy within 3 months before initiation of study treatment.
10. Use of strong cytochrome P450 isoform 3A inhibitors and inducers and drugs metabolized by cytochrome P450 isoform 3A, cytochrome P450 isoform 2B6, and cytochrome P450 isoform 1A2, and are identified as narrow therapeutic drugs within 7 days or 3 half-lives, whichever is longer, prior to initiation of study treatment
11. Adverse events from prior anticancer therapy that have not resolved to Grade ≤1, except for alopecia.
12. Prior autologous stem cell transplant within 6 months prior to the initiation of study treatment.
13. Prior allogeneic stem cell transplant within 6 months prior to the initiation of study treatment or with any evidence of active graft versus host disease or requirement for immunosuppressants within 28 days prior to the initiation of study treatment.
14. Clinically significant active infection (eg, pneumonia).
15. Major surgical procedure within 4 weeks prior to the initiation of study treatment.
16. Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
17. Pregnant (positive serum beta human chorionic gonadotropin test) or lactating women.
18. New York Heart Association Class II or greater congestive heart failure.
19. Congenital long QT syndrome or correct QT interval using Fridericia's formula (QTcF) >480 msec
20. Current use of medication known to cause QT prolongation or Torsades de Pointes
21. History of myocardial infarction or unstable angina within 6 months prior to the initiation of study treatment.
22. History of stroke or transient ischemic attack within 6 months prior to the initiation of study treatment.
23. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease.
24. Treatment in a clinical study within 30 days prior to the initiation of study treatment.
25. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Adverse Events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | From first dose to within 30 days after the last dose
  The safety and tolerability of HMPL-523 will be evaluated based on adverse events data.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From Cycle 1, Day 1, 5 min pre-dose 1st dose until Cycle 1, Day 28 8 hours post-dose.
  To Characterize the pharmacokinetic properties of HMPL-523 in patients with relapsed or refractory lymphoma
Area under the concentration-time curve in a selected time interval (AUC0-t) | From Cycle 1, Day 1, 5 min pre-dose 1st dose until Cycle 1, Day 28 8 hours post-dose.
  To characterize the pharmacokinetic properties of HMPL-523 in patients with relapsed or refractory lymphoma
Objective response rate (ORR) defined as the proportion of patients who have a CR or PR | From first dose to within 30 days after the last dose
  To evaluate the anti-tumor activity of HMPL-523 in patients with relapsed or refractory lymphoma according to: (1) Chronic Lymphocytic Leukemia (CLL) - modified International Workshop on CLL guidelines, (2) Waldenstrom's Macroglobulinemia (WM) - consensus of international workshops on WM, (3) Lymphomas other than CLL or WM: Lugano Response Criteria for Hodgkin and Non-Hodgkin's Lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Jayaprakash, MD, Study Director — Hutchmed
Locations (32):
- United States (8):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Innovative Clinical Research Institute, Downey, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Summit Medical Group, Florham Park, New Jersey
  - Clinical Research Alliance, New Hyde Park, New York
  - Leo Jenkins Cancer Center/ECU School of Medicine, Greenville, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
- Aarhus University Hospital, Aarhus, Denmark
- Finland (2):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Tampereen yliopistollinen sairaala, Tampere
- France (4):
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
- Italy (3):
  - Ospedale San Raffaele, Milan, Milano
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
- Poland (4):
  - KO-MED Centra Kliniczne, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego, Wroclaw
- Spain (10):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No